CLINICAL TRIAL: NCT07019844
Title: Addition of F18-Piflufolastat PET/CT to Cross-Sectional Imaging for the Staging and Management of Hepatocellular Carcinoma
Brief Title: PSMA PET for the Staging and Management of Hepatocellular Carcinoma
Status: Recruiting | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Miami VA Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: ONCC-006-23S; 1I01CX002654-01A1 (NIH); 1761959 (Other: VA Central Institutional Review Board Panel)
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Indeterminate Lesions Cohort (Diagnosis Focus): Participants in this cohort have liver lesions categorized as LI-RADS 3 or 4 based on standard imaging. The purpose of the PSMA PET/CT is to assist in the further characterization of these indeterminate nodules and support diagnosis of HCC or benign pathology.
- Treatment-Naïve Cohort (Staging Focus): This cohort includes participants with newly diagnosed HCC who have not yet received any locoregional or systemic therapy. PSMA PET/CT is performed to evaluate the extent of disease and detect potential intrahepatic or extrahepatic spread, contributing to improved staging accuracy.
- Post-Treatment Cohort (Treatment Response Focus): Participants in this cohort have previously undergone locoregional therapy (e.g., TACE, RFA, or ablation). PSMA PET/CT is used to assess residual or recurrent disease and help evaluate treatment response compared to standard imaging.

SUMMARY:
This prospective, single-center study evaluates the clinical utility of F18-Piflufolastat (PSMA) PET/CT when added to conventional cross-sectional imaging for patients with suspected or confirmed hepatocellular carcinoma (HCC). The study aims to determine whether PSMA PET/CT improves diagnostic accuracy for indeterminate liver lesions (LI-RADS 3 and 4), enhances staging precision in treatment-naïve patients, and provides more accurate assessment of treatment response in patients undergoing locoregional therapy (LRT). The goal is to assess how PSMA PET/CT may impact clinical decision-making, staging, and management of HCC across multiple stages of disease.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the most common primary liver cancer and a leading cause of cancer-related mortality worldwide. Accurate diagnosis, staging, and treatment response assessment are critical for optimal management of patients with HCC. However, conventional imaging modalities, such as contrast-enhanced CT and MRI, have limitations in characterizing indeterminate liver lesions and in detecting intrahepatic or extrahepatic disease, particularly in the context of post-treatment changes.

This prospective, single-center study investigates the added value of F18-Piflufolastat (PSMA) PET/CT in the evaluation and management of patients with suspected or confirmed HCC. PSMA (Prostate-Specific Membrane Antigen) is a cell surface protein that, while originally characterized in prostate cancer, has demonstrated overexpression in the neovasculature of a variety of solid tumors, including HCC. F18-Piflufolastat is a radiotracer that targets PSMA, allowing for enhanced molecular imaging.

Participants will undergo PSMA PET/CT imaging in addition to standard-of-care imaging (CT and/or MRI). The study is designed to address three primary clinical questions:

1. Diagnosis: Does the addition of PSMA PET/CT improve characterization of indeterminate liver lesions (e.g., LI-RADS 3 or 4)?
2. Staging: Can PSMA PET/CT improve the accuracy of disease staging in treatment-naïve patients by detecting intrahepatic or extrahepatic disease not visualized on conventional imaging?
3. Treatment Response: In patients who have undergone locoregional therapy (LRT), does PSMA PET/CT provide more precise assessment of viable tumor tissue compared to standard imaging? Data collected will include imaging results, histopathological confirmation when available, changes in clinical management prompted by PSMA PET/CT findings, and correlation with clinical outcomes. By evaluating the clinical utility of PSMA PET/CT across multiple phases of the disease course, this study aims to inform future diagnostic algorithms and treatment planning strategies in patients with HCC.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients age >18 years from the VA medical system
* Treatment-naïve patients with HCC with BCLC B or C disease

Exclusion Criteria:

* Patients with renal dysfunction or contrast allergy that precludes contrast enhanced cross sectional imaging
* Patients with presence of active primary malignancy other than HCC and non-melanoma skin cancer in the past 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will recruit 90 Veterans from the VHA with HCC, and no non-Veteran participants. This will include 30 participants with LR-3 and 4 lesions detected during surveillance (Aim 1), 30 treatment naïve participants towards Aim 2, and 30 treatment experienced participants for Aim 3. In addition, 10 participants out of the 60 who are recruited for aims 2 and 3 are projected to have indeterminate nodules, increasing the number of participants with indeterminate nodules to 40. West Palm Beach and Orlando VA patients who are evaluated at the Miami VA, will be approached for study recruitment. These Veterans will continue to be co-managed by the Miami VA and the local VA teams after undergoing treatment in Miami.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
1: Change in Diagnostic Classification of Indeterminate Lesions (LI-RADS 3/4) After PSMA PET/CT; 2: Change in Clinical Staging in Treatment-Naïve Patients; 3: Change in Assessment of Treatment Response Following Locoregional Therapy | 1: Within 30 days of PET/CT imaging; 2: Within 30 days of PET/CT imaging; 3: Within 30 days of post-treatment imaging
  1. Proportion of patients with LI-RADS 3/4 lesions whose diagnostic classification is revised (i.e., confirmed as HCC or benign) based on F18-Piflufolastat PET/CT findings, as compared to standard imaging alone. Final diagnosis will be based on histopathology (if available) or multidisciplinary tumor board consensus;
  2. Number and percentage of treatment-naïve patients whose disease stage is upstaged or down-staged after PSMA PET/CT imaging, relative to standard imaging, according to modified BCLC or AJCC staging guidelines;
  3. Difference in tumor viability classification based on PSMA PET/CT vs. standard imaging using mRECIST or LI-RADS treatment response criteria. Correlation with histopathologic or clinical follow-up will be evaluated where available.

SECONDARY OUTCOMES:
1: Change in Clinical Management Based on PSMA PET/CT Findings; 2: Change in Clinical Staging in Treatment-Naïve Patients; 3: Change in Assessment of Treatment Response Following Locoregional Therapy | 1: Within 30 days of PET/CT imaging; 2: Within 30 days of PET/CT imaging; 3: Within 30 days of post-treatment imaging
  1. Proportion of patients with LI-RADS 3/4 lesions whose diagnostic classification is revised (i.e., confirmed as HCC or benign) based on F18-Piflufolastat PET/CT findings, as compared to standard imaging alone. Final diagnosis will be based on histopathology (if available) or multidisciplinary tumor board consensus;
  2. Number and percentage of treatment-naïve patients whose disease stage is upstaged or downstaged after PSMA PET/CT imaging, relative to standard imaging, according to modified BCLC or AJCC staging guidelines;
  3. Difference in tumor viability classification based on PSMA PET/CT vs. standard imaging using mRECIST or LI-RADS treatment response criteria. Correlation with histopathologic or clinical follow-up will be evaluated where available.

OTHER OUTCOMES:
1: Inter-reader Agreement on PSMA PET/CT Interpretation; 2: Correlation Between PSMA Uptake and Histopathologic Features | 1: Within 30 days of imaging; 2: Up to 90 days post-imaging (when surgical specimens are available)
  1. Agreement between independent nuclear medicine readers on lesion characterization and treatment response using standardized reporting criteria (e.g., kappa statistics);
  2. Quantitative PET uptake metrics (SUVmax, SUVmean) will be correlated with histologic markers of tumor grade, vascular invasion, and PSMA expression, when pathology samples are available.

CONTACTS AND LOCATIONS:
Overall Officials: Binu V John, MD MPH, Principal Investigator — Miami VA Healthcare System, Miami, FL
Locations (1):
- Miami VA Healthcare System, Miami, FL, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
The United States Department of Veterans Affairs (VA) places legal restrictions on access to Veterans' healthcare data, including identifying and sensitive patient information. The analytic datasets used in this study were not permitted to leave the VA firewall without data-use agreement. This limitation is consistent with those of other studies based on VA data. However, VA data are freely available to researchers behind the VA firewall with an approved VA study protocol. For more information, please visit https://www.virec.research.va.gov or contact the VA Information Resource Center (VIReC) at Virec@Va.gov.

REFERENCES:
- [Background] John BV, Aubuchon S, Dahman B, Konjeti VR, Heuman D, Hubert J, Thomas S, Deng Y, Solomon C, Sundaram LT, Love E, Singal AG, Tatum JL. Addition of [18 F]Fluorodeoxyglucose Positron Emission Tomography With Computed Tomography to Cross-Sectional Imaging Improves Staging and Alters Management in Hepatocellular Carcinoma. Liver Transpl. 2020 Jun;26(6):774-784. doi: 10.1002/lt.25743. Epub 2020 May 8. PMID 32128966